CLINICAL TRIAL: NCT03187249
Title: Intervention Strategy in Chronic Obstructive Pulmonary Disease With Anxiety and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1304404B
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; Anxiety; Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy; Psychotherapy, Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Behavioral Therapy (Experimental): receive cognitive-behavioral therapy for 12 weeks
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Pulmonary Rehabilitation Therapy (Experimental): receive pulmonary rehabilitation therapy for 12 weeks
  Interventions: Behavioral: Pulmonary Rehabilitation Therapy
- Combined Therapy (Experimental): receive both cognitive-behavioral therapy and pulmonary rehabilitation therapy for 12 weeks
  Interventions: Behavioral: Combined Therapy
- Regular Therapy (No Intervention): receive regular therapy for chronic obstructive pulmonary disease

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 12 weeks cognitive-behavioral lessons, once a week
  Arms: Cognitive Behavioral Therapy
Behavioral: Pulmonary Rehabilitation Therapy — 12 weeks pulmonary rehabilitation exercise
  Arms: Pulmonary Rehabilitation Therapy
Behavioral: Combined Therapy — cognitive-behavioral lessons and pulmonary rehabilitation exercise for 12 weeks
  Arms: Combined Therapy

SUMMARY:
Anxiety and depression have negative effect on outcomes of chronic obstructive pulmonary disease (COPD). Intervention strategy including behavioral-cognitive therapy and pulmonary rehabilitation are promising in improving life quality, disease symptom and outcomes. But there's not standard algorithm in China so far. The study aims to compare the effectiveness of these interventions and develop an intervention algorithm of anxiety and depression in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD patients with mild or moderate anxiety and depression

Exclusion Criteria:

* Patients with bronchial asthma or other severe pulmonary diseases or having received pulmonary surgery in 6 months
* Patients with tumor history during past 5 years
* Patients with COPD exacerbations during past 4 weeks
* Participants in clinical trials
* Patients in pregnancy or breastfeeding
* Patients unable to complete questionaire independently
* Patients older than 80 years old
* Patients receiving long-term domiciliary oxygen therapy

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 12 weeks
  total score

SECONDARY OUTCOMES:
moderate and severe COPD exacerbations | 3 years
  total times
modified British medical research council score | 3 years
  total score
COPD assessment test score | 3 years
  total score

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided